CLINICAL TRIAL: NCT03325881
Title: A Phase 3, Randomized, Double-blind, Multicenter, Placebo-controlled, Fixed-Dose, Efficacy, and Safety Study of SHP465 in Children Aged 6-12 Years With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Efficacy and Safety of SHP465 at 6.25 mg in the Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in Children Aged 6-12 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP465-309
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Results first posted 2019-08-13 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; Hyperactivity; SHP465
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHP465 (Experimental): Participants will be randomized to receive SHP465 capsule 6.25 milligram (mg) orally once daily for 4 weeks.
  Interventions: Drug: SHP465
- Placebo (Placebo Comparator): Participant will receive placebo matching to SHP465 capsule orally once daily for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHP465 — SHP465 capsule 6.25 mg orally once daily for 4 weeks
  Arms: SHP465
Drug: Placebo — Placebo matching to SHP465 capsule orally once daily for 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHP465 at 6.25 mg in the treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in children aged 6-12 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female aged 6-12 years inclusive at the time of consent.
* Participant's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (as applicable) by the participant.
* Participant must meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (any subtype).
* Participant who is a female and of child-bearing potential must not be pregnant and agree to comply with any applicable contraceptive requirements.
* Participant has an ADHD-RS-5 Child, Home Version Total Score of greater than or equal to (>=) 28 and Clinical Global Impression - Severity of Illness (CGI-S) score >=4 at baseline (Visit 2). Participant is currently not on ADHD therapy, or is not completely satisfied with their current ADHD therapy.

Exclusion Criteria:

* Participant is required or anticipated to take medications that have central nervous system effects or affect performance. Stable use of bronchodilator inhalers is not exclusionary.
* Participant has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the participant.
* Participant has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
* Participant has failed to fully respond, based on investigator judgment, to an adequate course of amphetamine therapy.
* Participant has a known family history of sudden cardiac death or ventricular arrhythmia.
* Participant has a blood pressure measurement >=95th percentile for age, sex, and height at screening (Visit 1) and/or baseline (Visit 2).
* Participant has a height less than or equal to (<=) 5th percentile for age and sex at screening (Visit 1) or baseline (Visit 2).
* Participant has a weight <=5th percentile for age and sex at screening (Visit 1) or baseline (Visit 2).
* Participant has a known history of symptomatic cardiovascular disease, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, or other serious cardiac conditions placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Participant has a history of seizures (other than infantile febrile seizures).
* Participant is taking any medication that is excluded per the protocol.
* Participant had any clinically significant ECG or clinical laboratory abnormalities at the screening (Visit 1) or baseline visit (Visit 2).
* Participant has current abnormal thyroid function, defined as abnormal thyroid-stimulating hormone and thyroxine at the screening or baseline visit. Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Participant has a current, controlled (requiring medication or therapy) or uncontrolled, comorbid psychiatric disorder.
* Participant is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of or currently demonstrating suicidal ideation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2017-12-09 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (41):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - PEWMD, PA, ARCSM, PLLC, PRP, Inc., Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Riverside Medical Clinic, Riverside, California
  - Peninsula Research Associates - CRN, Rolling Hills, California
  - Care Research Center, Doral, Florida
  - Power MD Clinical Research Institute, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Acevedo Medical Group, Miami, Florida
  - Pharmacology Research, LLC, Miami, Florida
  - Scientific Clinical Research Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Clinical Associates of Orlando, Llc, Orlando, Florida
  - GA Psychiatric Services, LLC., Atlanta, Georgia
  - Buford Family Practice, Buford, Georgia
  - One Health Research Clinic, Inc., Norcross, Georgia
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Advanced Clinical Research Inc., Meridian, Idaho
  - Conventions Psychiatry and Counseling, Naperville, Illinois
  - Pedia Research, LLC, Evansville, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Neuroscientific Insights, Rockville, Maryland
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - St Charles Psychiatric Associates, Saint Charles, Missouri
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Pediatric Associates, Mt. Pleasant, South Carolina
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - El Campo Clinical Trials, El Campo, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Children's Clinic, League City, Texas
  - University of Texas, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - VA South Psychiatric & Family Services, Petersburg, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Mid-Columbia Research, Richland, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mattingly G, Arnold V, Yan B, Yu M, Robertson B. A Phase 3, Randomized Double-Blind Study of the Efficacy and Safety of Low-Dose SHP465 Mixed Amphetamine Salts Extended-Release in Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2020 Nov;30(9):549-557. doi: 10.1089/cap.2020.0005. Epub 2020 Oct 13. PMID 33185468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 43 study centers in the United States between 09 December 2017 (first participant first visit) and 07 June 2018 (last participant last visit).
Pre-assignment Details: A total of 124 participants were screened, of them 89 were randomized and 88 received the treatment. Out of them, 83 participants completed the study.
Groups:
- Placebo: Participants received placebo matched to SHP465 capsule orally once daily for 4 weeks.
- SHP465: Participants received 6.25 milligrams (mg) SHP465 capsule orally once daily for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | SHP465
Started | 44 | 45
Treated | 43 | 45
Completed | 41 | 42
Not Completed | 3 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants in the randomized set who took at least 1 dose of investigational product.
Groups:
- SHP465: Participants received 6.25 mg SHP465 capsule orally once daily for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | SHP465 | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.8 (2.03) | 8.8 (2.20) | 8.8 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 29 | 27 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 20 | 37
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28 | 30 | 58
  Race: Black or African American | 10 | 11 | 21
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Other | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale-5 (ADHD-RS-5) Total Score at Week 4
Description: Clinician administered ADHD-RS-5, child, home version total score were analyzed. ADHD-RS-5 consisted of 18 items designed to reflect current symptomatology of ADHD based on diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) criteria. Each item was scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items were grouped into 2 subscales: hyperactivity or impulsivity (9 items) and inattentiveness (9 items). Higher total scores indicated higher impairment and lower scores indicated no impairment. Least square (LS) mean was calculated based on restricted maximum likelihood (REML) method of estimation and utilized an unstructured covariance type.
Time Frame: Baseline, Week 4
Population: Full analysis set consisted of all participants in the safety set who had baseline ADHD-RS-5 total score and at least 1 postdose ADHD-RS-5 total score. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 40 | 42
Score on a scale | -9.7 [-13.2 to -6.2] | -11.6 [-15.0 to -8.2]
Statistical Analysis 1: Comparison: Placebo vs SHP465; Number of participants with SHP465 was compared with placebo using the linear mixed-effects model for repeated measures (MMRM) that included treatment group, nominal visit, age group, interaction of the treatment group with the visits as factors, baseline ADHD-RS5 total score as a covariate and an adjustment for the interaction of the baseline ADHD-RS-5 Total Score with the visit; Test type: Superiority; p = 0.451, Mixed-effects model for repeated measure; Difference in LS Mean = -1.9, 95% CI 2-sided [-6.8 to 3.1], Standard Error of Mean 2.48

2. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Week 4
Description: CGI scale was measured to rate the overall improvement of a participants condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). LS mean was calculated based on restricted maximum likelihood (REML) method of estimation and utilized an unstructured covariance type.
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 40 | 42
Score on a scale | 3.3 [3.0 to 3.6] | 3.2 [2.9 to 3.5]
Statistical Analysis 1: Comparison: Placebo vs SHP465; Number of participants with SHP465 was compared with placebo using the mixed effects model for repeated measures (MMRM) that includes treatment group, nominal visit, age group,interaction of the treatment group with the visit as factors, baseline CGI-S as a covariate and an adjustment for the interaction of the baseline CGI-S with the visit; Test type: Superiority; p = 0.597, Mixed-effects model for repeated measure; Difference in LS mean = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.20

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that start or deteriorate on or after the date of the first dose of investigational product and no later than 3 days following the last dose of investigational product.
Time Frame: From start of study drug administration up to follow-up (Week 5)
Population: Safety set consisted of all participants in the randomized set who as taken at least 1 dose of investigator product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
Participants | 7 | 11

4. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs Were Reported as Adverse Event (AE)
Description: Vital sign assessments included systolic and diastolic blood pressure and pulse. Participants with clinically significant deviations from baseline values which are deemed clinically significant in the opinion of the investigator were considered as AE's. An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: From start of study drug administration up to follow-up (Week 5)
Population: Safety set consisted of all participants in the randomized set who taken at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participant received placebo matched to SHP465 capsule orally once daily for 4 weeks.
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
Participants
  Number of participants with secondary hypertension | 1 | 0
  Number of participants with Tachycardia | 1 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Change in Clinical Laboratory Test Results Assessed by the Investigator
Description: Clinical laboratory tests included biochemistry, endocrinology, hematology and urinalysis. The investigator assessed out-of-range clinical laboratory values for clinical significance, if the value(s) were not clinically significant or clinically significant.
Time Frame: From start of study drug administration up to follow-up (Week 5)
Population: Safety set consisted of all participants in the randomized set who taken at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Assessed by the Investigator
Description: Participants with clinically significant deviations from baseline values which are deemed clinically significant in the opinion of the investigator were considered in 12-lead ECG and reported.
Time Frame: From start of study drug administration up to follow-up (Week 5)
Population: Safety set consisted of all participants in the randomized set who taken at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Quality of Sleep Assessed by Post Sleep Questionnaire (PSQ) at Baseline and Week 4
Description: The PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collected data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. Participants analyzed for number of times woke up per night category were only the participants who responded as yes for the woke up during the night category in this outcome measure.
Time Frame: Baseline, Week 4
Population: Safety set consisted of all participants in the randomized set who taken at least 1 dose of investigational product. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 42
Participants
  Baseline: Woke up during the night - Yes | 20 | 14
  Baseline: Woke up during the night - No | 23 | 28
  Week 4: Woke up during the night - Yes: number analyzed (Participants) | 40 | 42
  Week 4: Woke up during the night - Yes | 13 | 11
  Week 4: Woke up during the night - No: number analyzed (Participants) | 40 | 42
  Week 4: Woke up during the night - No | 27 | 31
  Baseline: Number of times woke up per night = 0: number analyzed (Participants) | 20 | 14
  Baseline: Number of times woke up per night = 0 | 0 | 1
  Baseline: Number of times woke up per night = 1: number analyzed (Participants) | 20 | 14
  Baseline: Number of times woke up per night = 1 | 12 | 6
  Baseline: Number of times woke up per night = 2: number analyzed (Participants) | 20 | 14
  Baseline: Number of times woke up per night = 2 | 8 | 6
  Baseline: Number of times woke up per night = 3: number analyzed (Participants) | 20 | 14
  Baseline: Number of times woke up per night = 3 | 0 | 1
  Baseline: Number of times woke up per night = 4: number analyzed (Participants) | 20 | 14
  Baseline: Number of times woke up per night = 4 | 0 | 0
  Baseline: Number of times woke up per night >= 5: number analyzed (Participants) | 20 | 14
  Baseline: Number of times woke up per night >= 5 | 0 | 0
  Week 4: Number of times woke up per night = 0: number analyzed (Participants) | 13 | 11
  Week 4: Number of times woke up per night = 0 | 0 | 1
  Week 4: Number of times woke up per night = 1: number analyzed (Participants) | 13 | 11
  Week 4: Number of times woke up per night = 1 | 8 | 8
  Week 4: Number of times woke up per night = 2: number analyzed (Participants) | 13 | 11
  Week 4: Number of times woke up per night = 2 | 5 | 1
  Week 4: Number of times woke up per night = 3: number analyzed (Participants) | 13 | 11
  Week 4: Number of times woke up per night = 3 | 0 | 0
  Week 4: Number of times woke up per night = 4: number analyzed (Participants) | 13 | 11
  Week 4: Number of times woke up per night = 4 | 0 | 1
  Week 4: Number of times woke up per night >= 5: number analyzed (Participants) | 13 | 11
  Week 4: Number of times woke up per night >= 5 | 0 | 0
  Baseline: Was the past week a typical week - Yes | 39 | 36
  Baseline: Was the past week a typical week - No | 4 | 6
  Week 4: Was the past week a typical week - Yes: number analyzed (Participants) | 40 | 42
  Week 4: Was the past week a typical week - Yes | 36 | 36
  Week 4: Was the past week a typical week - No: number analyzed (Participants) | 40 | 42
  Week 4: Was the past week a typical week - No | 4 | 6
  Baseline: Past week was not typical - Vacation: number analyzed (Participants) | 4 | 6
  Baseline: Past week was not typical - Vacation | 2 | 2
  Baseline: Past week was not typical - School break: number analyzed (Participants) | 4 | 6
  Baseline: Past week was not typical - School break | 1 | 2
  Baseline: Past week was not typical - Friend house: number analyzed (Participants) | 4 | 6
  Baseline: Past week was not typical - Friend house | 0 | 0
  Baseline: Past week was not typical - ill: number analyzed (Participants) | 4 | 6
  Baseline: Past week was not typical - ill | 0 | 0
  Baseline: Past week was not typical - other: number analyzed (Participants) | 4 | 6
  Baseline: Past week was not typical - other | 1 | 2
  Week 4: Past week was not typical - Vacation: number analyzed (Participants) | 4 | 6
  Week 4: Past week was not typical - Vacation | 0 | 0
  Week 4: Past week was not typical - School break: number analyzed (Participants) | 4 | 6
  Week 4: Past week was not typical - School break | 3 | 3
  Week 4: Past week was not typical - Friend house: number analyzed (Participants) | 4 | 6
  Week 4: Past week was not typical - Friend house | 0 | 0
  Week 4: Past week was not typical - ill: number analyzed (Participants) | 4 | 6
  Week 4: Past week was not typical - ill | 0 | 1
  Week 4: Past week was not typical - other: number analyzed (Participants) | 4 | 6
  Week 4: Past week was not typical - other | 1 | 2
  Baseline : Overall quality - Better than usual: number analyzed (Participants) | 8 | 9
  Baseline : Overall quality - Better than usual | 0 | 1
  Baseline: Overall quality - Same as usual: number analyzed (Participants) | 8 | 9
  Baseline: Overall quality - Same as usual | 6 | 7
  Baseline: Overall quality - Worse than usual: number analyzed (Participants) | 8 | 9
  Baseline: Overall quality - Worse than usual | 2 | 1
  Week 4: Overall quality - Better than usual: number analyzed (Participants) | 5 | 11
  Week 4: Overall quality - Better than usual | 1 | 2
  Week 4: Overall quality - Same as usual: number analyzed (Participants) | 5 | 11
  Week 4: Overall quality - Same as usual | 4 | 7
  Week 4: Overall quality - Worse than usual: number analyzed (Participants) | 5 | 11
  Week 4: Overall quality - Worse than usual | 0 | 2

8. Secondary Outcome: Change From Baseline in Length of Time Awake Per Night and Length of Time to Fall Asleep Per Night Assessed by PSQ at Week 4
Description: The PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collected data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week.
Time Frame: Baseline, Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
minutes
  Baseline: Length of Time to fall asleep per night: number analyzed (Participants) | 43 | 42
  Baseline: Length of Time to fall asleep per night | 27.0 (20.25) | 27.2 (21.51)
  Week 4: Length of Time to fall asleep per night: number analyzed (Participants) | 40 | 42
  Week 4: Length of Time to fall asleep per night | 19.3 (16.13) | 21.0 (14.35)
  Baseline: Length of Time awake per night: number analyzed (Participants) | 20 | 14
  Baseline: Length of Time awake per night | 12.4 (8.41) | 8.0 (7.63)
  Week 4: Length of Time awake per night: number analyzed (Participants) | 12 | 11
  Week 4: Length of Time awake per night | 8.9 (5.18) | 15.1 (17.01)

9. Secondary Outcome: Change From Baseline in Length of Time Sleeping Per Night Assessed by PSQ at Week 4
Description: as for outcome 8
Time Frame: Baseline, Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
hours
  Baseline: number analyzed (Participants) | 43 | 42
  Baseline | 8.9 (1.20) | 8.8 (1.22)
  Week 4: number analyzed (Participants) | 40 | 42
  Week 4 | 9.1 (1.34) | 8.9 (1.16)

10. Secondary Outcome: Total Sleep Disturbance Score of Children's Sleep Habits Questionnaire (CSHQ ) at Week 4
Description: The CSHQ is a validated, retrospective, parent-reported sleep screening tool. The questionnaire consists of 35 items that yield a TSD score, as well as 8 subscale scores, including bedtime resistance, sleep duration, parasomnias, sleep disordered breathing, night wakings, daytime sleepiness, sleep anxiety, and sleep onset delay. Parents were asked to think of a recent "typical" week of their child's sleep and to indicate how often sleep disturbance behaviors occurred. A 3-point scale was used for rating: "usually" if the sleep behavior occurs 5 to 7 times per week, "sometimes" for 2 to 4 times per week, and "rarely" for once or not at all during the week. The TSD score, which is the sum of all responses, included all items of the 8 subscales, but consisted of only 33 items because two on the bedtime resistance and sleep anxiety subscales were identical (range: 0, 99). A negative value indicates less sleep disturbance.
Time Frame: Week 4
Population: Safety set consisted of all participants in the randomized set who took at least 1 dose of SHP465. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 41 | 41
Units on scale | 42.7 (9.36) | 42.8 (9.17)

11. Secondary Outcome: Number of Participants With a Positive Response in Columbia-suicide Severity Rating Scale (C-SSRS) at Week 4
Description: C-SSRS was a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The number of participants with clinical significant change in suicidal ideation and suicidal behavior were reported.
Time Frame: Week 4
Population: Safety set consisted of all participants in the randomized set who took at least 1 dose of investigational product. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 43 | 45
Participants
  Suicidal Ideation: number analyzed (Participants) | 41 | 42
  Suicidal Ideation | 0 | 0
  Suicidal Behavior: number analyzed (Participants) | 41 | 42
  Suicidal Behavior | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Week 5)
Description: Safety analysis was analysed for the safety population (88 participants) and not for the enrolled population as in participant flow (89 participants).
Groups:
- SHP465: Participants received 6.25 milligram (mg) of SHP465 capsule orally once daily for 4 weeks.
Arm/Group | Placebo | SHP465
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45
Other Adverse Events (participants affected / at risk) | 3/43 | 2/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | SHP465 (N=45)
Headache (Nervous system disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03325881/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03325881/SAP_001.pdf